CLINICAL TRIAL: NCT05137002
Title: A Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Multiple Dose Strengths of CIN-107 as Compared to Placebo After 8 Weeks of Treatment in Patients With Uncontrolled Hypertension
Brief Title: A Study of CIN-107 in Patients With Uncontrolled Hypertension
Acronym: HALO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CinCor Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN-107-124
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Uncontrolled Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CIN-107 0.5 mg (Experimental): Remain on background anti-hypersensitive regimen for 8 weeks. After 8 weeks, patient will receive the highest dose of CIN-107 (2 mg) and discontinue their background antihypertensive agent(s) for 4 weeks
  Interventions: Drug: CIN-107
- CIN-107 1 mg (Experimental): Remain on background anti-hypersensitive regimen for 8 weeks. After 8 weeks, patient will receive the highest dose of CIN-107 (2 mg) and discontinue their background antihypertensive agent(s) for 4 weeks
  Interventions: Drug: CIN-107
- CIN-107 2 mg (Experimental): Remain on background anti-hypersensitive regimen for 8 weeks. After 8 weeks, patient may remain on CIN-107 (2 mg) and discontinue their background antihypertensive agent(s) for 4 weeks or withdraw study participation depending on BP control
  Interventions: Drug: CIN-107
- Placebo (Placebo Comparator): Remain on background anti-hypersensitive regimen for 8 weeks. After 8 weeks, patient will receive the highest dose of CIN-107 (2mg) and discontinue their background antihypertensive agent(s) for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CIN-107 — CIN-107 tablets by mouth once daily
  Other Names: Baxdrostat
  Arms: CIN-107 0.5 mg; CIN-107 1 mg; CIN-107 2 mg
Drug: Placebo — Placebo tablets by mouth once daily
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, multicenter study to evaluate the efficacy and safety of multiple dose strengths of baxdrostat (also called CIN-107) in the treatment of patients with uncontrolled hypertension. The primary objective was to demonstrate that treatment with baxdrostat for 8 weeks would lower the systolic blood pressure (SBP) in patients who were hypertensive despite taking one or two anti-hypertensive medications.

Participants were assigned to take placebo or baxdrostat once per day for 8 weeks while they continued taking the regular anti-hypertensive medications. At the end of the 8-week period, qualified patients could participate in Part II of the study and receive 2 mg baxdrostat for 4 weeks while they discontinued taking the background anti-hypertensive medication.

ELIGIBILITY:
Inclusion Criteria:

* Is on a stable regimen of background antihypertensive agent(s) for at least 8 weeks and would be considered a candidate for an additional antihypertensive agent at the time of screening ;
* Has a mean seated systolic blood pressure (SBP) ≥ 140 mmHg or ≥ 130 mmHg if diabetic;
* Demonstrates ability to be adherent to the study drug and their anti-hypertensive medication during a run-in period
* If taking an SGLT2 inhibitor, the regimen must be stable for at least 8 weeks prior to randomization; and
* Agrees to comply with the contraception and reproduction restrictions of the study;

Exclusion Criteria:

* Has a mean seated systolic blood pressure (SBP) ≥180 mmHG;
* Has a body mass index (BMI) >50 kg/m2;
* Is using alpha or beta blockers for any primary indication other than systemic hypertension (eg, migraine headache);
* Is not willing or not able to discontinue an MRA or potassium sparing diuretic as part of an existing antihypertensive regimen;
* Has documented estimated eGFR <30 mL/min/1.73m2;
* Has known and documented New York Heart Association stage III or IV chronic heart failure;
* Has had a stroke, transient ischemic attack, hypertensive encephalopathy, acute coronary syndrome, or hospitalization for heart failure within 6 months before screening;
* Major cardiac surgery within 6 months before Screening;
* Has chronic permanent atrial fibrillation;
* Has uncontrolled diabetes with glycated hemoglobin >10% at Screening;
* Has planned dialysis or kidney transplantation planned during the course of the study;
* Prior solid organ transplant and/or cell transplants;
* Sodium <130 mEq/L;
* Potassium <3.5 mEq/L;
* Potassium >5 mEq/L;
* White blood cell count >15 × E9/L or absolute neutrophil count <1 × E9/L at Screening;
* Is positive for HIV antibody, hepatitis C virus RNA, or hepatitis B surface antigen;
* Has typical consumption of ≥14 alcoholic drinks weekly;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - CinCor Site 27, Saraland, Alabama
  - CinCor Site 35, Tucson, Arizona
  - CinCor Site 69, Encinitas, California
  - CinCor Site 6, Lincoln, California
  - CinCor Site 20, Los Angeles, California
  - CinCor Site 70, Lynwood, California
  - CinCor Site 36, Northridge, California
  - CinCor Site 29, Oceanside, California
  - CinCor Site 46, Panorama City, California
  - CinCor Site 47, San Dimas, California
  - CinCor Site 49, Santa Ana, California
  - CinCor Site 52, West Hills, California
  - CinCor Site 57, Denver, Colorado
  - CinCor Site 31, Waterbury, Connecticut
  - CinCor Site 18, Clearwater, Florida
  - CinCor Site 41, Cooper City, Florida
  - CinCor Site 28, Homestead, Florida
  - CinCor Site 9, Jupiter, Florida
  - CinCor Site 1, Lake Worth, Florida
  - CinCor Site 12, Miami, Florida
  - CinCor Site 54, Miami, Florida
  - CinCor Site 13, Miami, Florida
  - CinCor Site 17, Miami, Florida
  - CinCor Site 16, Tampa, Florida
  - CinCor Site 34, Winter Haven, Florida
  - CinCor Site 14, Buford, Georgia
  - CinCor Site 33, Addison, Illinois
  - CinCor Site 40, Chicago, Illinois
  - CinCor Site 42, Gurnee, Illinois
  - CinCor Site 50, Morton, Illinois
  - CinCor Site 72, Brownsburg, Indiana
  - CinCor Site 63, West Des Moines, Iowa
  - CinCor Site 7, Lexington, Kentucky
  - CinCor Site 21, Louisville, Kentucky
  - CinCor Site 30, Marrero, Louisiana
  - CinCor Site 59, Metairie, Louisiana
  - CinCor Site 19, New Orleans, Louisiana
  - CinCor Site 25, Shreveport, Louisiana
  - CinCor Site 38, Elkridge, Maryland
  - CinCor Site 22, Troy, Michigan
  - CinCor Site 64, Olive Branch, Mississippi
  - CinCor Site 11, Brooklyn, New York
  - CinCor Site 65, Staten Island, New York
  - CinCor Site 15, Cincinnati, Ohio
  - CinCor Site 24, Columbus, Ohio
  - CinCor Site 4, Dayton, Ohio
  - CinCor Site 43, Oklahoma City, Oklahoma
  - CinCor Site 60, Chattanooga, Tennessee
  - CinCor Site 48, Austin, Texas
  - CinCor Site 32, Carrollton, Texas
  - CinCor Site 68, Dallas, Texas
  - CinCor Site 61, Georgetown, Texas
  - CinCor Site 55, Houston, Texas
  - CinCor Site 3, Houston, Texas
  - CinCor Site 58, Katy, Texas
  - CinCor Site 62, Lampasas, Texas
  - CinCor Site 26, McAllen, Texas
  - CinCor Site 53, San Antonio, Texas
  - CinCor Site 10, Sugar Land, Texas
  - CinCor Site 45, Salt Lake City, Utah
  - CinCor Site 2, Manassas, Virginia
  - CinCor Site 5, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A Run-In Period up to 4 weeks before randomization, to confirm the patient's adherence to their background antihypertensive medication(s) and placebo was done. A total of 631 patients were screened for the study, of which 382 (60.5%) patients failed the screening. Two hundred forty-nine patients were randomized to 1 of the 4 treatment groups.
Groups:
- Placebo: Placebo: Placebo tablets by mouth once daily. IMP is taken as add-on while remaining on background anti-hypersensitive regimen for 8 weeks (Part I).
  After 8 weeks, patients will receive the highest dose of CIN-107 (2mg) and discontinue their background antihypertensive agent(s) for 4 weeks (Part II)
- CIN-107 0.5 mg: CIN-107: (0.5mg) CIN-107 tablets by mouth once daily. IMP is taken as add-on while remaining on background anti-hypersensitive regimen for 8 weeks (Part I).
  After 8 weeks, patients will receive the highest dose of CIN-107 (2 mg) and discontinue their background antihypertensive agent(s) for 4 weeks (Part II)
- CIN-107 1 mg: CIN-107: (1mg) CIN-107 tablets by mouth once daily. IMP is taken as add-on while remaining on background anti-hypersensitive regimen for 8 weeks (Part I).
  After 8 weeks, patients will receive the highest dose of CIN-107 (2 mg) and discontinue their background antihypertensive agent(s) for 4 weeks (Part II)
- CIN-107 2 mg: CIN-107: (2mg) CIN-107 tablets by mouth once daily. IMP is taken as add-on while remaining on background anti-hypersensitive regimen for 8 weeks (Part I).
  After 8 weeks, patients may remain on CIN-107 (2 mg) and discontinue their background antihypertensive agent(s) for 4 weeks (Part II) or withdraw study participation depending on BP control
- Part II - CIN-107 2mg: CIN-107: (2mg) CIN-107 tablets by mouth once daily.
  After 8 weeks, patients may switch to or remain on 2mg CIN-107 and discontinue their background antihypertensive agent(s) for 4 weeks (Part II).
Period: Part I (8 Weeks)
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg | Part II - CIN-107 2mg
Started | 64 | 63 | 62 | 60 | 0
Completed | 60 | 55 | 58 | 54 | 0
Not Completed | 4 | 8 | 4 | 6 | 0
Period: Part II (4 Weeks)
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg | Part II - CIN-107 2mg
Started | 0 | 0 | 0 | 0 | 213 (A total of 227 participants completed Part I, but 14 (1 of 0.5mg CIN-107 Part I, 1 of 1mg CIN-107 Part I, and 12 of 2mg CIN-107 Part I) of these participants did not enter Part II, 213 participants entered Part II.)
Completed | 0 | 0 | 0 | 0 | 201
Not Completed | 0 | 0 | 0 | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg | Total
Number analyzed (Participants) | 64 | 63 | 62 | 60 | 249
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 37 | 37 | 41 | 155
  >=65 years | 24 | 26 | 25 | 19 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.61) | 59.9 (10.85) | 61.2 (10.69) | 59.2 (11.88) | 60.2 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 28 | 37 | 30 | 132
  Male | 27 | 35 | 25 | 30 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 39 | 28 | 35 | 133
  Not Hispanic or Latino | 33 | 24 | 34 | 25 | 116
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 17 | 14 | 15 | 14 | 60
  White | 46 | 48 | 43 | 44 | 181
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 64 | 63 | 62 | 60 | 249
Seated SBP [Mean (Standard Deviation); unit: mmHg] | 147.9 (9.33) | 146.3 (8.60) | 147.0 (9.07) | 146.3 (7.83) | 146.9 (8.71)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Seated Systolic BP (SBP)
Description: The primary efficacy endpoint was the change from baseline in mean seated SBP after 8 weeks of treatment in patients with uncontrolled HTN (Part 1).
Time Frame: 8 weeks
Population: mITT Population - Four subjects (1, 2, 1 subjects from Placebo, 0.5mg CIN 107, and 2mg CIN 107, respectively) discontinued Part 1 early, but had their early termination (ET) visits within Week 8/Visit 6 analysis visit window.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg
Number analyzed (Participants) | 61 | 57 | 58 | 55
mmHg | -16.6 (1.58) | -17.0 (1.63) | -16.0 (1.62) | -19.8 (1.67)

2. Secondary Outcome: Change From Baseline in Mean Seated Diastolic BP (DBP)
Description: The change from baseline in mean seated DBP with CIN-107 compared to placebo after 8 weeks of treatment (Part 1)
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg
Number analyzed (Participants) | 61 | 57 | 58 | 55
mmHg | -5.9 (1.17) | -5.8 (1.20) | -5.0 (1.19) | -5.4 (1.23)

3. Secondary Outcome: Change From Baseline in 24-hour Urine Aldosterone
Description: The change from baseline in 24-hour urine aldosterone levels with CIN 107 compared to placebo after 8 weeks of treatment (Part 1)
Time Frame: 8 weeks
Population: mITT population - Two subjects discontinued Part 1 early, but had their ET measures taken within Week8/Visit 6 analysis visit window: 1 from Placebo and 1 from 0.5mg. In addition, 7 subjects completed Part 1 but either did not have baseline measure or did not have Week 8/Visit 6 measure: 2, 2, 3 subjects from Placebo, 0.5mg CIN 107, and 1mg CIN 107, respectively.
Measure: Least Squares Mean (Standard Error); unit: ng/g
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg
Number analyzed (Participants) | 59 | 54 | 55 | 54
ng/g | -19.90 (29.183) | -114.16 (31.305) | -140.45 (29.999) | -121.64 (30.760)

4. Secondary Outcome: Change From Baseline in 24-hour Serum Aldosterone
Description: The change from baseline in 24-hour serum aldosterone levels with CIN 107 compared to placebo after 8 weeks of treatment (Part 1)
Time Frame: 8 weeks
Population: mITT population - Four subjects discontinued Part 1 early, but had their ET measures taken within Week8/Visit 6 analysis visit window: 1, 2, 1 subjects from Placebo, 0.5mg CIN 107, and 2mg CIN 107, respectively. In addition, 13 subjects completed Part 1 but either did not have baseline measure or did not have Week 8/Visit 6 measure: 4, 6, 3 subjects from Placebo, 1mg CIN 107, and 2mg CIN 107, respectively.
Measure: Least Squares Mean (Standard Error); unit: ng/dL
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg
Number analyzed (Participants) | 57 | 57 | 52 | 52
ng/dL | -0.70 (0.490) | -2.76 (0.493) | -2.95 (0.508) | -2.92 (0.515)

5. Secondary Outcome: Percentage of Patients Achieving a Mean Seated SBP <130 mmHg
Description: The percentage of patients achieving a mean seated SBP <130 mmHg ("responders") with CIN-107 compared to placebo after 8 weeks of treatment (Part 1; Weeks 1 to 8)
Time Frame: 8 weeks
Population: mITT population - Patients without a Week 8/Visit 6 systolic blood pressure measure were considered non-responders. So, if a subject was in the mITT Population but discontinued the study early or if SBP measure was unavailable at Week 8, then they were considered non responders and still contributed to the total number of participants used in analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg
Number analyzed (Participants) | 64 | 63 | 62 | 60
Participants | 36 | 36 | 33 | 43

6. Secondary Outcome: Change From Baseline in 24-hour Urine Renin
Description: The change from baseline in 24-hour urine renin levels with CIN-107 compared to placebo after 8 weeks of treatment (Part 1)
Time Frame: 8 weeks
Population: mITT population - The 24 hour urine renin pharmacodynamic analyte was added in later, with protocol v3.0. Only subjects who had this measured at baseline are included in overall number of participants analyzed.
Measure: Least Squares Mean (Standard Error); unit: ng/day
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg
Number analyzed (Participants) | 5 | 4 | 10 | 4
ng/day | -20.08 (16.584) | -6.54 (15.739) | -5.74 (10.703) | 4.11 (17.930)

7. Secondary Outcome: Change From Baseline in 24-hour Serum Renin
Description: The change from baseline in 24-hour serum renin levels with CIN-107 compared to placebo after 8 weeks of treatment (Part 1)
Time Frame: 8 weeks
Population: mITT population - The 24 hour serum renin pharmacodynamic analyte was added in later, with protocol v3.0. Only subjects who had this measured at baseline are included in overall number of participants analyzed.
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg
Number analyzed (Participants) | 5 | 2 | 10 | 4
ng/L | 92.902 (144.3969) | 63.565 (195.0495) | 88.041 (91.2996) | -140.961 (151.5431)

ADVERSE EVENTS:
Time Frame: Part I - AEs during the 8-week treatment period Part II - AEs during the following 4-week treatment period
Groups:
- Placebo: CIN-107: CIN-107 tablets by mouth once daily. Remain on background anti-hypersensitive regimen for 8 weeks (part I).
  After 8 weeks, patients will receive the highest dose of CIN-107 (2mg) and discontinue their background antihypertensive agent(s) for 4 weeks (part II)
- CIN-107 0.5 mg; CIN-107 1 mg: CIN-107: CIN-107 tablets by mouth once daily. Remain on background anti-hypersensitive regimen for 8 weeks (part I).
  After 8 weeks, patients will receive the highest dose of CIN-107 (2 mg) and discontinue their background antihypertensive agent(s) for 4 weeks (part II)
- CIN-107 2 mg: CIN-107: CIN-107 tablets by mouth once daily. Remain on background anti-hypersensitive regimen for 8 weeks (part I).
  After 8 weeks, patients may remain on CIN-107 (2 mg) and discontinue their background antihypertensive agent(s) for 4 weeks (part II) or withdraw study participation depending on BP control
- Part II - CIN-107 2 mg: CIN-107: (2mg) CIN-107 tablets by mouth once daily and discontinue their background anti-hypertensive agent(s) for 4 weeks (Part II).
Arm/Group | Placebo | CIN-107 0.5 mg | CIN-107 1 mg | CIN-107 2 mg | Part II - CIN-107 2 mg
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63 | 0/62 | 1/60 | 0/213
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/63 | 1/62 | 1/60 | 3/213
Other Adverse Events (participants affected / at risk) | 5/64 | 8/63 | 6/62 | 3/60 | 6/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | CIN-107 0.5 mg (N=63) | CIN-107 1 mg (N=62) | CIN-107 2 mg (N=60) | Part II - CIN-107 2 mg (N=213)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | CIN-107 0.5 mg (N=63) | CIN-107 1 mg (N=62) | CIN-107 2 mg (N=60) | Part II - CIN-107 2 mg (N=213)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 5 (5) | 3 (3) | 6 (6)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo for up to 90 days.

DOCUMENTS (2):
  • Study Protocol (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT05137002/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT05137002/SAP_001.pdf